CLINICAL TRIAL: NCT05404594
Title: Multimodal Approach to the Ontogenesis of Nociception in Very Preterm and Term Infants
Acronym: NOCI-Prem
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 7256
Record Dates: First submitted 2022-02-21; First posted 2022-06-03 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Procedural Pain; Pre-Term; Venipuncture
Keywords: Very preterm infants; Development of nociception; Cortical hemodynamic responses; Pain indicators; Gender; Maternal voice; Oxytocin
MeSH Terms: conditions — Pain, Procedural; Premature Birth; Coitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Very preterm infant (Experimental): Preterm infant below 33 weeks of GA
  Interventions: Behavioral: Maternal vocal contact
- Full term neonate (Active Comparator): Term neonate from a gestational age of 37 weeks.
  Interventions: Behavioral: Maternal vocal contact

INTERVENTIONS:
Behavioral: Maternal vocal contact — Two consecutive venipuncture (order randomly balanced) within a short period of time will be realized with and without the presence of the mother talking/singing to her VPI infant.
  In this intervention group, the mother will be supported to talk or to sing to her infants during before and during the venipuncture.

SUMMARY:
The management of pain related to venipuncture remains insufficient in very preterm infants (VPI. The separation between the mother (father) and her(his) child can aggravate the short-term painful experience of the newborn. Accurate diagnosis and treatment of pain is necessary to preserve the well-being and brain development of VPI. A better understanding of the development of pain pathways and the cortical integration of nociceptive messages is essential to reach this goal.

ELIGIBILITY:
Inclusion Criteria:

* Experimental group: VPIs of gestational age less than or equal to 33 weeks on the day of birth and hospitalized in the neonatal intermediate care unit or the neonatal intensive care unit of the Neonatal department of the Hautepierre Hospital (Strasbourg University Hospital)

  * Control group: Healthy full-term babies (> 37 weeks gestational age) hospitalized in the maternity ward of Strasbourg University Hospital
  * Consent obtained from both parents
  * Subject affiliated to a social health insurance plan.

Exclusion Criteria:

* - Any malformation known before inclusion
* Cerebral lesions discovered on cerebral ultrasound performed as part of the standard management of newborns (Intra-Ventricular Hemorrhages of grade III or IV of the Papile classification, Periventricular Leucomalacia)
* Unstable clinical status according to the investigator's judgment
* Expected transfer of the child to another hospital before the term of 40 weeks PMAs.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-07-17 (Actual); Primary Completion 2023-04-17 (Estimated); Study Completion 2023-04-17 (Estimated)

PRIMARY OUTCOMES:
The cortical hemodynamic response profile | During a venipuncture (needed for the standard care of the infants) and realized around 30 (+/- 2) weeks PMAs in VPI
  The measurements will be performed using receiver and transmitter optodes to measure the variations of oxy and deoxyhemoglobin in the cerebral cortex below the optodes. The optodes will be placed in the primary and secondary somatosensory areas, and in other cortical areas (nociceptive pathway and control areas) using the EEG 10-20 classification. The data set will be collected over a basal period, a stimulation period and a post-stimulation period. Response patterns will be analyzed by mixed models and compared in VPIs in the different APM groups and with term neonates. A typical response associates an increase in oxyhemoglobin (Hb02) with a concomitant stability or decrease in deoxyhemoglobin (HHb).
The cortical hemodynamic response profile | During a venipuncture at 34 (+/-2) weeks PMAs in VPI
  The measurements will be performed using receiver and transmitter optodes to measure the variations of oxy and deoxyhemoglobin in the cerebral cortex below the optodes. The optodes will be placed in the primary and secondary somatosensory areas, and in other cortical areas (nociceptive pathway and control areas) using the EEG 10-20 classification. The data set will be collected over a basal period, a stimulation period and a post-stimulation period. Response patterns will be analyzed by mixed models and compared in VPIs in the different APM groups and with term neonates. A typical response associates an increase in oxyhemoglobin (Hb02) with a concomitant stability or decrease in deoxyhemoglobin (HHb).
The cortical hemodynamic response profile | During a venipuncture at 40 (+/-2) weeks PMAs in VPI
  The measurements will be performed using receiver and transmitter optodes to measure the variations of oxy and deoxyhemoglobin in the cerebral cortex below the optodes. The optodes will be placed in the primary and secondary somatosensory areas, and in other cortical areas (nociceptive pathway and control areas) using the EEG 10-20 classification. The data set will be collected over a basal period, a stimulation period and a post-stimulation period. Response patterns will be analyzed by mixed models and compared in VPIs in the different APM groups and with term neonates. A typical response associates an increase in oxyhemoglobin (Hb02) with a concomitant stability or decrease in deoxyhemoglobin (HHb).
The cortical hemodynamic response profile | During a venipuncture at 2 to 3 days of life in term neonates
  The measurements will be performed using receiver and transmitter optodes to measure the variations of oxy and deoxyhemoglobin in the cerebral cortex below the optodes. The optodes will be placed in the primary and secondary somatosensory areas, and in other cortical areas (nociceptive pathway and control areas) using the EEG 10-20 classification. The data set will be collected over a basal period, a stimulation period and a post-stimulation period. Response patterns will be analyzed by mixed models and compared in VPIs in the different APM groups and with term neonates. A typical response associates an increase in oxyhemoglobin (Hb02) with a concomitant stability or decrease in deoxyhemoglobin (HHb).

SECONDARY OUTCOMES:
Comparison of the hemodynamic response profiles and salivary oxytocin levels | During a venipuncture (needed for the standard care of the infants) and realized around 30 (+/- 2) weeks PMAs in VPI
  Comparison of the hemodynamic response profiles and salivary oxytocin levels during 2 consecutive venipunctures, without and with the addition of the maternal voice as a supplementary non-pharmacological pain strategies
Comparison of the hemodynamic response profiles and salivary oxytocin levels | During a venipuncture at 34 (+/-2) weeks PMAs in VPI
  Comparison of the hemodynamic response profiles and salivary oxytocin levels during 2 consecutive venipunctures, without and with the addition of the maternal voice as a supplementary non-pharmacological pain strategies
Comparison of the hemodynamic response profiles and salivary oxytocin levels | During a venipuncture at 40 (+/-2) weeks PMAs in VPI
  Comparison of the hemodynamic response profiles and salivary oxytocin levels during 2 consecutive venipunctures, without and with the addition of the maternal voice as a supplementary non-pharmacological pain strategies
Comparison of the hemodynamic response profiles and salivary oxytocin levels | During a venipuncture at 2 to 3 days of life in term neonates
  Comparison of the hemodynamic response profiles and salivary oxytocin levels during 2 consecutive venipunctures, without and with the addition of the maternal voice as a supplementary non-pharmacological pain strategies
Analysis of the impact on the responses of maternal separation | During a venipuncture (needed for the standard care of the infants) and realized around 30 (+/- 2) weeks PMAs in VPI
  Analysis of the impact on the responses of maternal separation determined by the absence of early skin-to-skin contact (in the VPI < 3 days of life and in the term newborn < 2 hours of life).
Analysis of the impact on the responses of maternal separation | During a venipuncture at 34 (+/-2) weeks PMAs in VPI
  Analysis of the impact on the responses of maternal separation determined by the absence of early skin-to-skin contact (in the VPI < 3 days of life and in the term newborn < 2 hours of life).
Analysis of the impact on the responses of maternal separation | During a venipuncture at 40 (+/-2) weeks PMAs in VPI
  Analysis of the impact on the responses of maternal separation determined by the absence of early skin-to-skin contact (in the VPI < 3 days of life and in the term newborn < 2 hours of life).
Analysis of the impact on the responses of maternal separation | During a venipuncture at 2 to 3 days of life in term neonates
  Analysis of the impact on the responses of maternal separation determined by the absence of early skin-to-skin contact (in the VPI < 3 days of life and in the term newborn < 2 hours of life).
Comparison of the response profiles according to the sex | During a venipuncture (needed for the standard care of the infants) and realized around 30 (+/- 2) weeks PMAs in VPI
  Comparison of the response profiles obtained in females and males
Comparison of the response profiles according to the sex | During a venipuncture at 34 (+/-2) weeks PMAs in VPI
  Comparison of the response profiles obtained in females and males
Comparison of the response profiles according to the sex | During a venipuncture at 40 (+/-2) weeks PMAs in VPI
  Comparison of the response profiles obtained in females and males
Comparison of the response profiles according to the sex | During a venipuncture at 2 to 3 days of life in term neonates
  Comparison of the response profiles obtained in females and males
Comparison of conduction velocities of small caliber nociceptive fibers | During a venipuncture (needed for the standard care of the infants) and realized around 30 (+/- 2) weeks PMAs in VPI
  Comparison of conduction velocities of small caliber nociceptive fibers measured by evoked potentials, in response to non-painful cold stimulation in the VPIs of different APMs groups.
Comparison of conduction velocities of small caliber nociceptive fibers | During a venipuncture at 34 (+/-2) weeks PMAs in VPI
  Comparison of conduction velocities of small caliber nociceptive fibers measured by evoked potentials, in response to non-painful cold stimulation in the VPIs of different APMs groups.
Comparison of conduction velocities of small caliber nociceptive fibers | During a venipuncture at 40 (+/-2) weeks PMAs in VPI
  Comparison of conduction velocities of small caliber nociceptive fibers measured by evoked potentials, in response to non-painful cold stimulation in the VPIs of different APMs groups.
Comparison of conduction velocities of small caliber nociceptive fibers | During a venipuncture at 2 to 3 days of life in term neonates
  Comparison of conduction velocities of small caliber nociceptive fibers measured by evoked potentials, in response to non-painful cold stimulation in the VPIs of different APMs groups.
Correlational analyses by APM group | During a venipuncture (needed for the standard care of the infants) and realized around 30 (+/- 2) weeks PMAs in VPI
  Correlational analyses, by APM group, between the different pain indicators in response to stimulation
Correlational analyses by APM group | During a venipuncture at 34 (+/-2) weeks PMAs in VPI
  Correlational analyses, by APM group, between the different pain indicators in response to stimulation
Correlational analyses by APM group | During a venipuncture at 40 (+/-2) weeks PMAs in VPI
  Correlational analyses, by APM group, between the different pain indicators in response to stimulation
Correlational analyses by APM group | During a venipuncture at 2 to 3 days of life in term neonates
  Correlational analyses, by APM group, between the different pain indicators in response to stimulation
Facial pain behavior | During a venipuncture (needed for the standard care of the infants) and realized around 30 (+/- 2) weeks PMAs in VPI
  Facial pain behavior with the Neonatal Facial Coding System
Facial pain behavior | During a venipuncture at 34 (+/-2) weeks PMAs in VPI
  Facial pain behavior with the Neonatal Facial Coding System
Facial pain behavior | During a venipuncture at 40 (+/-2) weeks PMAs in VPI
  Facial pain behavior with the Neonatal Facial Coding System
Facial pain behavior | During a venipuncture at 2 to 3 days of life in term neonates
  Facial pain behavior with the Neonatal Facial Coding System
Pain index | During a venipuncture (needed for the standard care of the infants) and realized around 30 (+/- 2) weeks PMAs in VPI
  Pain index assessing the sympathetic and parasympathetic system
Pain index | During a venipuncture at 34 (+/-2) weeks PMAs in VPI
  Pain index assessing the sympathetic and parasympathetic system
Pain index | During a venipuncture at 40 (+/-2) weeks PMAs in VPI
  Pain index assessing the sympathetic and parasympathetic system
Pain index | During a venipuncture at 2 to 3 days of life in term neonates
  Pain index assessing the sympathetic and parasympathetic system
Cortical evoked potentials | During a venipuncture (needed for the standard care of the infants) and realized around 30 (+/- 2) weeks PMAs in VPI
  Cortical evoked potentials in Cz according to EEG 10:20 classification
Cortical evoked potentials | During a venipuncture at 34 (+/-2) weeks PMAs in VPI
  Cortical evoked potentials in Cz according to EEG 10:20 classification
Cortical evoked potentials | During a venipuncture at 40 (+/-2) weeks PMAs in VPI
  Cortical evoked potentials in Cz according to EEG 10:20 classification
Cortical evoked potentials | During a venipuncture at 2 to 3 days of life in term neonates
  Cortical evoked potentials in Cz according to EEG 10:20 classification

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pédiatrie - Hôpital d'Hautepierre, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No